CLINICAL TRIAL: NCT06127199
Title: A Single Arm, Open-Label Pivotal Contraceptive Efficacy Study of Ovaprene
Brief Title: Contraceptive Efficacy Study of Ovaprene
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daré Bioscience, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DR-OVP-002
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Contraception
Keywords: Device; Non-hormonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Ovaprene (Experimental)
  Interventions: Device: Ovaprene

INTERVENTIONS:
Device: Ovaprene — Non-hormonal intravaginal ring

SUMMARY:
This will be a multi-center, single arm, open-label study of Ovaprene, a non-hormonal intravaginal ring, to investigate the contraceptive effectiveness, safety and acceptability of Ovaprene.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active people assigned female at birth, at risk for pregnancy and desiring contraception.
* General good health, by subject history and per investigator judgement
* Age 18 through 40 years, inclusive; approximately 66 subjects >35 years old at visit 2 will be the Enrolled-Eligible Population
* In a relationship with a person assigned male at birth who meets eligibility criteria below.

  --At least 18 years old, not known to be subfertile or infertile
* Have regular menstrual cycles (when not on hormonal contraception) with a usual length of 21 to 35 days, without heave bleeding that lasts longer than 5 days
* Be willing to stop their current method of contraception (with the exception of condoms) before Visit 2. Participants must experience at least one subsequent menstrual bleed before inserting Ovaprene. Participants using injectable contraception must be at least 9 months post their last dose at screening and have experienced at least 2 subsequent regular menstrual bleeds that were part of cycles of 21-35 days. After stopping their current method of contraception, subjects must either abstain fro vaginal sex or use condoms before inserting their first Ovaprene
* Not be actively desiring pregnancy for at least 13 months and be willing to accept an unknown risk of pregnancy
* Expect to engage in at least 4 acts of heterosexual vaginal intercourse per cycle during the study.
* Be willing to only use Ovaprene as the sole method of contraception over the course of the study
* Agree not to participate in any other clinical trials during the course of the study
* Be willing and able to comply with study procedures and to return to the clinic for scheduled follow-up visits
* Microbiota/innate immunity and colposcopy subsets only:

  * Be willing to avoid vaginal sex and using tampons and other intravaginal products for 48 hours prior to clinic visits; and be willing to comply with subset procedures

Exclusion Criteria:

* Currently pregnant and/or have a positive urine pregnancy test at screening.
* Have an allergy to the ingredients in Ovaprene
* Have a history of toxic shock syndrome
* Have a history of hereditary hemochromatosis
* Be breastfeeding an infant
* Have a history suggestive of infertility, defined as any of the following: known history of ectopic pregnancy or other fertility problem; sterilization/permanent contraception; endometriosis or hospitalization for pelvic inflammatory disease (PID) unless subject has had a subsequent spontaneous intrauterine pregnancy; or use of medications that could cause subfertility such as gonadotropin-releasing hormone agonists
* Currently have postcoital bleeding
* Have contraindications to pregnancy (medical condition) or chronic use of medications contraindicated in pregnancy
* Have a history of clinically significant uterine prolapse, cystocele, or rectocele that has required surgical intervention or pessary use
* Positive human immunodeficiency virus (HIV) test at screening
* Have exclusionary results on human papilloma virus (HPV) screening/cytology (subjects>/=21 years old) at screening or require treatment or follow-up for an abnormal Pap smear or HPV test that would be needed during the study.
* Have had a vaginal or cervical biopsy within 1 month or vaginal surgery within the 3 months prior to screening
* Known current drug or alcohol abuse which, in the opinion of the investigator, could impact study compliance
* Have previously been included in the Enrolled-Eligible Population
* Is a direct employee or immediate family member of the Sponsor company, site Investigators or study staff
* Have taken any investigational drug or used any investigational device within the 30 days prior to screening
* Have a history of any severe acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation or study treatment administration or could interfere with the interpretation of trial results
* Microbiota/innate immunity subset only:

  --systemic use in the last 2 weeks prior to screening or anticipated use during the study of antibiotics (other than those used to treat urinary tract infection (UTI), candidiasis, or bacterial vaginosis(BV) diagnosed at Visit 1) or antivirals;
* If male partner has or is suspected to have had an HIV infection or other sexually transmitted infection
* if male partner has a known sensitivity or allergy to the ingredients in Ovaprene
* If male partner has previously participated in this study or has taken any investigational drug or used any investigational device within 30 days prior to the female subject's screening
* If the male partner has a history of any severe acute or chronic medical or psychiatric condition that could increase the risk associated with trial participation or could interfere with the interpretation of trial results.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 656 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Determination of pregnancy rate | 12 months
  Measurement of number of pregnancies over 13 menstrual cycles (13-cycle Pearl Index)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Mauck, MD, Study Director — Daré Bioscience, Inc.
Locations (27):
- United States (27):
  - Precision Trials AZ, Phoenix, Arizona
  - MomDoc Women's Health Research, Scottsdale, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Essential Health Access (Berkeley), Berkeley, California
  - Essential Access Health, Los Angeles, California
  - Amicis Research Center, Newhall, California
  - University of California at Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Praetorian Pharmaceutical Research, LLC, Marrero, Louisiana
  - The Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Rutgers Medical Center, Newark, New Jersey
  - Columbia University, New York, New York
  - Einstein College of Medicine, The Bronx, New York
  - Carolina Women's Research and Wellness Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Penn Obstetric Gynecology Associates, Philadelphia, Pennsylvania
  - Magee-Women's Hospital, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Seattle Clinical Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Final decision on what will be shared has not yet been determined.